CLINICAL TRIAL: NCT04871594
Title: A Phase 1b Trial in Stage II-III Urothelial Cancer to Explore Pre-operative Immunotherapy
Brief Title: Pre-operative Immunotherapy in Stage II-III Urothelial Cancer
Acronym: TURANDOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: 4SC AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21TUR
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label phase 1b clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab monotherapy (Experimental): Day 1: nivolumab 240 mg Day 22: nivolumab 240 mg Day 43: nivolumab 240 mg
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — On day 1, 22, and 43 240mg
  Other Names: Opdivo

SUMMARY:
This is a phase 1b feasibility study of pre-operative immunotherapy in PD-L1 positive resectable stage II-III urothelial cancer patients. This study can be adapted or expanded based on the results obtained.

DETAILED DESCRIPTION:
This is a phase 1b feasibility study of pre-operative immunotherapy in PD-L1 positive resectable stage II-III urothelial cancer patients.

Urothelial cancer patients will be included that are diagnosed with either:

* cT2-4aN0M0 OR
* cT1-4aN1-3M0

PD-L1 status will be determined. When PD-L1 CPS is ≥10%, patients will be treated with three cycles nivolumab 240 mg, q3wk, on day 1, 22, 43.

The primary endpoint is feasibility of pre-operative nivolumab in PD-L1 positive resectable stage II-III urothelial cancer patients.

After surgery, patients attend study visits at day 8 and at day 29. Their final study visit for physical examination and laboratory testing is at day 57 (+/- 7 days), which is scheduled to anticipate late-onset adverse events. 90 days postoperative, surgical complications according to the Clavien-dindo classification will be evaluated. Thereafter, patients will be followed according to standard clinical guidelines. Tumor biopsies/material preservation is required at baseline and during surgery.

Main secondary endpoints are:

* To identify pathological complete response rates of nivolumab in PD-L1 positive resectable stage II-III urothelial cancer patients
* To describe immune-related grade 3/4 and all grade toxicities
* To describe RFS and OS
* Translational: Effects of immunotherapy on the tumor microenvironment based on RNA signatures and changes in immune infiltrates between baseline and resection.

ELIGIBILITY:
Inclusion criteria:

1. Willing and able to provide informed consent
2. Age ≥ 18 years
3. Resectable muscle-invasive UC (upper urinary tract allowed), defined as:

   * cT2-4aN0M0 OR
   * cT1-4aN1-3M0
4. World Health Organization (WHO) performance Status 0 or 1.
5. Urothelial cancer is the dominant histology (>70%).
6. Formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks from diagnostic TUR available (or equivalent FFPE tumor specimens for upper tract tumors; at least two biopsy cores available).
7. PD-L1 status must be determined using the 22C3 pharmDx test. Combined positivity score (CPS) must be >10.
8. Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥1.0x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, GFR>30 ml/min as per Cockcroft-Gault formula, AST ≤ 1.5 x ULN, ALT ≤1.5 x ULN, Bilirubin ≤1.5 X ULN
9. Negative pregnancy test (βHCG in blood or urine) for female patients of childbearing potential within 2 weeks prior to Day 1 Cycle 1.
10. Highly effective contraception for both male and female subjects if the risk of conception exists. Female patients of childbearing potential must comply with contraception methods as requested by the study protocol.

Exclusion criteria:

1. Subjects with active autoimmune disease in the past 2 years. Patients with diabetes mellitus, properly controlled hypothyroidism or hyperthyroidism, vitiligo, psoriasis or other mild skin disease can still be included.
2. Documented history of severe autoimmune disease (e.g. inflammatory bowel disease, myasthenia gravis).
3. Prior CTLA-4 or PD-1/PD-L1-targeting immunotherapy.
4. Known history of Human Immunodeficiency Virus infection or tuberculosis, or other active infection requiring therapy at the time of inclusion.
5. Positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
6. Underlying medical conditions that, in the investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of adverse events
7. Medical condition requiring the use of immunosuppressive medications, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) will be allowed.
8. Use of other investigational drugs before study drug administration
9. Malignancy, other than urothelial cancer, in the previous 2 years, with a high chance of recurrence (estimated >10%). Patients with low risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
10. Pregnant and lactating female patients.
11. Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
12. Severe infections within 2 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
13. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, unstable arrhythmias and unstable angina.
14. Previous intravenous chemotherapy for bladder cancer. Prior low-dose sensitizing chemotherapy used for combined modality treatment, or radiation alone, is allowed if patients have recurred after an initial response. Patients with residual disease after (chemo)radiation for bladder cancer are not eligible.
15. Patients in whom use of a colon segment for urinary diversion is planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of pre-operative nivolumab in PD-L1 positive resectable stage II-III urothelial cancer patients | At 12 weeks
  Percentage of patients that underwent surgery within 12 weeks after study start will be assessed

SECONDARY OUTCOMES:
Pathological complete response rates of nivolumab in PD-L1 positive resectable stage II-III urothelial cancer patients | At 12 weeks
  Efficacy of nivolumab in PD-L1 positive resectable stage II-III urothelial cancer patients, assessed by the percentage of pathological complete response rate after cystectomy according to pathological response criteria
Toxicity of pre-operative nivolumab | From first inusion untill 100 days after the last infusion with nivolumab
  All grade toxicities and immune-related toxicity of grade 3-4
Relapse free survival and overall survival | From first infusion untill 3 years postoperative
  During follow-up, every 6 months untill 3 years postoperative, relapse free survival will be evaluated. Overall survival will be evaluated by phone calls
Monitor peri-surgical complications | From surgery untill 90 days after surgery
  Peri-operative complications and morbidity will be graded according to the Clavien-Dindo classification
Translational: effects of nivolumab on the tumor microenvironment | At 12 weeks
  Resistance mechanisms are explored by comparing immune (cell) infiltrates in responders and nonresponders in pre- and post treatment tissue [Multiplex immunohistochemistry, RNA seq]

CONTACTS AND LOCATIONS:
Overall Officials: M.S. van der Heijden, Dr., Principal Investigator — The Netherlands Cancer Institute
Locations (2):
- Netherlands (2):
  - Antoni van Leeuwenhoek ziekenhuis, Amsterdam
  - Radboud Universitair Medisch Centrum, Nijmegen